CLINICAL TRIAL: NCT03861325
Title: Insuffisance Gastro-intestinale Aiguë Translocation Microbienne Chez Les Patients en Choc Septique : Une étude Pilote
Brief Title: Acute Intestinal Failure in Critically Ill Patients and Microbial Translocation
Acronym: IGA-TM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02192-53; 2018-A02192-53 (Other: ANSM)
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2020-12

CONDITIONS: Septic Shock
Keywords: acute gut failure
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis of the investigators is that patients with septic shock in ICU have acute intestinal insufficiency favoring subclinical microbial translocation, which is the consequence of alterations of the epithelium, and is accompanied by qualitative and quantitative changes in the gut microbiota.

The primary objective is to determine the incidence of microbial translocation by measuring 16S rDNA and 18S rDNA plasma levels in a patient population with septic shock.

Secondary objectives are:

* Describe the kinetics of markers of intestinal insufficiency (I-FABP / zonulin) over time (at admission, 12 hours after admission, one day, two day, three days and seven day after admission).
* Study the correlation between the titer of I-FABP, zonulin, 16srDNA, 18srDNA and the stages of acute gastrointestinal insufficiency (AGF).
* Establish correlations between the microorganisms of the intestinal microbiota and the bacteria involved in microbial translocation.
* Study the possible correlations between the 16SrDNA levels and the other bacterial markers (sCD14, LBP).
* Describe the evolution of the composition and the diversity of the gut microbiota in the first 7 days of septic shock

DETAILED DESCRIPTION:
All eligible patients admitted for septic shock in resuscitation at Nimes will be included in the study, after verification of inclusion and non-inclusion criteria and with their agreement.

This is an observational study with no impact on the quality of care provided. All study data will be entered into an electronic CRF (e-CRF) directly or from the paper version of the scorecard.

The entry into the e-CRF is controlled and formatted to prohibit the input of out-of-bounds or outliers. In case of modification of data entry, traceability and monitoring of activities is ensured. An electronic signature committing the responsibility of the investigator of each center will allow the validation of the visit and the e-CRF.

Only those persons participating in the research project and identified will have access to the software allowing this entry: Redcap.

Redcap software that allows you to generate electronic CRFs (e-CRF), electronically capture data, manage it and restore it. It also makes it possible to follow the progress of studies in terms of data entry and to manage them. It is open source software that is extensible, modular and based on international standards.

Redcap software allows:

* Data entry, validation and annotation by clinicians and research associates
* Data extraction, filtering and analysis by investigators
* Study management by study coordinators
* Monitoring, auditing, configuration and reporting by administrators The electronic observation notebook creation software is hosted on a website within the CHU of Nîmes. Access to this application is secure and is via a password. Data collected through this software is backed up daily on a secure network. The network is connected to the internet, the access is protected by a firewall.

The clinical data of the study will be stored on a specific directory of the server. Only the network administrators and the authorized persons of the clinical research unit of the medical information department can have access to this directory.

IT arrangements made to enforce the confidentiality commitment

* The technical resources are located in the IT department whose access is controlled and secure.
* The data is stored on a server hosted in a secure room at the CHU Nîmes.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his / her representative has been informed about the implementation of the study, its objectives, its constraints, the rights of the patient and must have received the newsletter and no opposition of the study.
* The patient must be an affiliate or beneficiary of a health insurance plan.
* The patient is at least 18 years old.
* The patient has septic shock as defined by the 3rd International Conference for the definition of sepsis and septic shock

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under guardianship, under guardianship, or under the protection of justice
* The patient has already participated in this study
* The patient or his / her representative refuses to participate in the study
* The patient is pregnant, parturient or is breastfeeding
* The patient is a minor
* The patient is in therapeutic limitation or moribund
* The patient has undergone or is going to have scheduled or emergency digestive surgery
* The patient is HIV-positive
* The patient has Child C cirrhosis
* The patient has progressive digestive neoplasia, digestive lymphoma, chronic inflammatory bowel disease (Crohn's disease ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Describe the incidence of microbial translocation in critical illness by measuring 16S rDNA and 18S rDNA plasma levels in a patient population with septic shock | 7 days
  Plasma levels of circulating 16S rDNA and 18S rDNA will be measured at admission in ICU then 12 hours, 1 day, 2 days, 3 days and seven days later after admission.

SECONDARY OUTCOMES:
Describe the kinetics of markers of intestinal insufficiency by measuring I-FABP and Zonulin plasma levels | 7 days
  Plasma levels of I-FABP and Zonulin will be measured at admission in ICU then 12 hours, 1 day, 2 days, 3 days and seven days later after admission.
Study the correlation between the titer of I-FABP, zonulin, 16S rDNA, 18S rDNA and the stages of acute gastrointestinal insufficiency (AGF) | 7 days
  Plasma levels of 16S rDNA, 18S rDNA, I-FABP and Zonulin will be measured at admission in ICU then 12 hours, 1 day, 2 days, 3 days and seven days later after admission and stages of AGF will be evaluated at the same time.
Establish correlations between the microorganisms of the intestinal microbiota and the bacteria involved in microbila translocation | 7 days
  the results of the qualitative analysis of the microbiota will be compared with the results of the classic microbiological samples taken on admission to the intensive care unit
Study the possible correlations between the 16SrDNA plasma levels and the other bacterial markers (plasma levels of sCD14, LBP) | 7 days
  Plasma levels of 16S rDNA, sCD14 and LBP will be measured at admission in ICU then 12 hours, 1 day, 2 days, 3 days and seven days later after admission.
Perform a qualitative and quantitative analysis of the intestinal microbiota at admission to intensive care and after 7 days from a stool sample taken on admission to intensive care on the seventh day after admission | 7 days
  The metagenomic analysis of the gut microbiota is based on the high-throughput sequencing of all bacteria in a stool sample by targeting the 16S rRNA genes. The first step of this technique is to PCR amplify a 16S rDNA genomic target (eg V3-V4 regions) from stool sample DNA and to control the amplified sequences (called "libraries"). The second step consists in sequencing the libraries on a sequencing automaton. The bioinformatic analysis of the sequences consists of making a reference sequence library of the 16S rDNA target and aligning the sequences obtained with this database in order to establish lists of present organisms and taxonomic trees (OTU - operational taxonomic unit).

CONTACTS AND LOCATIONS:
Locations (1):
- Nimes University Hospital, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magnan C, Lancry T, Salipante F, Trusson R, Dunyach-Remy C, Roger C, Lefrant JY, Massanet P, Lavigne JP. Role of gut microbiota and bacterial translocation in acute intestinal injury and mortality in patients admitted in ICU for septic shock. Front Cell Infect Microbiol. 2023 Dec 18;13:1330900. doi: 10.3389/fcimb.2023.1330900. eCollection 2023. PMID 38179421